CLINICAL TRIAL: NCT03965520
Title: Exercise Test and Sequential Training Strategies in Peripheral Arterial Disease
Brief Title: Exercise Test and Sequential Training Strategies in PAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103-4837B
Record Dates: First submitted 2019-05-17; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; exercise training; local aerobic training
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual training (Active Comparator): exercise intensity arranged by cardiopulmonary exercise test results
  Interventions: Behavioral: exercise rehabilitation by near-infrared spectrometer
- Novel exercise training (Experimental): exercise intensity monitor by near-infrared spectrometer
  Interventions: Behavioral: exercise rehabilitation by near-infrared spectrometer

INTERVENTIONS:
Behavioral: exercise rehabilitation by near-infrared spectrometer — We adjust exercise intensity by the oxygen saturation change show in near-infrared spectrometer

SUMMARY:
Diabetic lower extremity disease, including peripheral vascular disease, peripheral neuropathy, foot ulcers, or leg amputation. Among them, peripheral arterial disease (PAD) is an important expression of systemic atherosclerosis. With the progress of the disease, impaired peripheral blood circulation will lead to many symptoms and signs, such as pain, paresthesia, and numbness.

In past studies show that regular exercise with moderate intensity may help to improve metabolism and hemodynamic characteristics of the individual. In addition, many studies have found that despite substantial organic changes in downstream tissue, exercise training can improve walking ability and aerobic capacity in patients with peripheral arterial disease.

To enhance exercise capacity in patients with PAD may involve redistribution of blood ﬂow from vascular beds with lower O 2 exchange rates towards exercising ischemic muscles, an increase in nutritive leg muscle blood ﬂow at the expense of regional shunting mechanisms, increased peripheral O 2 use during exercise attributable to more optimal distribution of leg blood ﬂow, and possible increased muscle capillary density and mitochondrial capacity.

Therefore, we tried to mimic local (leg) ischemic- reperfusion by systemic exercise, or to practice remote preconditioning effect by interval occlusion of the blood vessel in the upper arm which acquired ischemic preconditioning effect, and to improve local blood flow. Furthermore, the hemagglutination performance in PAD patients may also be used as an important indicator of cardiovascular disease.

DETAILED DESCRIPTION:
Diabetic lower extremity disease, including peripheral vascular disease, peripheral neuropathy, foot ulcers, or leg amputation. Among them, peripheral arterial disease (PAD) is an important expression of systemic atherosclerosis. With the progress of the disease, impaired peripheral blood circulation will lead to many symptoms and signs, such as pain, paresthesia, and numbness.

In past studies show that regular exercise with moderate intensity may help to improve metabolism and hemodynamic characteristics of the individual. In addition, many studies have found that despite substantial organic changes in downstream tissue, exercise training can improve walking ability and aerobic capacity in patients with peripheral arterial disease.

To enhance exercise capacity in patients with PAD may involve redistribution of blood ﬂow from vascular beds with lower O 2 exchange rates towards exercising ischemic muscles, an increase in nutritive leg muscle blood ﬂow at the expense of regional shunting mechanisms, increased peripheral O 2 use during exercise attributable to more optimal distribution of leg blood ﬂow, and possible increased muscle capillary density and mitochondrial capacity.

Therefore, we tried to mimic local (leg) ischemic- reperfusion by systemic exercise, or to practice remote preconditioning effect by interval occlusion of the blood vessel in the upper arm which acquired ischemic preconditioning effect, and to improve local blood flow. Furthermore, the hemagglutination performance in PAD patients may also be used as an important indicator of cardiovascular disease

ELIGIBILITY:
Inclusion Criteria:

* Ankle-brachial index <0.9

Exclusion Criteria:

* 1.<20 years old 2. There are other diseases or behavioral restrictions that prevent exercise training 3. Other exercise contraindications:

  1. unstable angina
  2. resting systolic blood pressure greater than 200 mmHg or diastolic blood pressure greater than 110 mmHg
  3. orthostatic blood pressure drop greater than 20 mmHg with symptoms
  4. Symptomatic severe aortic stenosis
  5. Acute systemic infection, accompanied by fever, body aches, or swollen lymph glands
  6. Uncontrolled cardiac dysrhythmias causing symptoms or hemodynamic compromise
  7. Uncontrolled symptomatic heart failure
  8. High-degree atrioventricular blocks
  9. Acute myocarditis or pericarditis
  10. Acute pulmonary embolus or pulmonary infarction
  11. a recent significant change in the resting electrocardiogram suggesting significant ischemia,
  12. recent myocardial infarction (within 2 d), or other acute cardiac events

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
physical fitness (peak oxygen consumption) | after 36 session exercise training, up to 12 weeks
  oxygen consumption in cc/min/kg measured by Carefusion(TM) during cardiopulmonary exercise test
physical fitness (exercise duration) | after 36 session exercise training, up to 12 weeks
  exercise duration in seconds measured during cardiopulmonary exercise test
physical fitness (walking distance) | after 36 session exercise training, up to 12 weeks
  walking distance in meters measured during six minutes walking test

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Medicine and Rehabilitation of Keelung Chang Gung Memorial hospital, Keelung, Taiwan